CLINICAL TRIAL: NCT02766205
Title: Prediction of Atrial Fibrillation in Patients With Embolic Stroke of Undetermined Source (AF-ESUS)
Brief Title: Prediction of AF in ESUS
Acronym: AF-ESUS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Thessaly (Other)
Collaborators: University of Lausanne (Other); University of Athens (Other)
Responsible Party: Principal Investigator, George Ntaios, MD, MSc (ESO Stroke Medicine), PhD, FESO, Assistant Professor of Internal Medicine, Medical School, University of Thessaly, Larissa University Hospital, University of Thessaly
Other Study IDs: WI211961
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: Embolic Stroke of Undetermined Source; Atrial fibrillation; prognostic score
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the proposed study is to identify predictors of covert atrial fibrillation (AF) in Embolic Stroke of Undetermined Source (ESUS) patients and develop a prognostic score for the identification of covert AF in this population.

DETAILED DESCRIPTION:
A new clinical entity termed Embolic Stroke of Undetermined Source (ESUS) was recently introduced by the Cryptogenic Stroke/ESUS International Working Group, which describes stroke patients for whom the source of embolism remains undetected despite thorough investigation; potential embolic sources include diseases of the mitral and aortic valves, the left cardiac chambers, the proximal cerebral arteries of the aortic arch and the venous system via paradoxical embolism. ESUS has been proposed as a potential therapeutic entity with a possible indication for anticoagulation, a hypothesis which is currently tested in two randomized controlled trials.

ESUS is defined as a visualized non-lacunar brain infarct in the absence of a) extracranial or intracranial atherosclerosis causing ≥50% luminal stenosis in arteries supplying the area of ischaemia, b) major-risk cardioembolic source, and c) any other specific cause of stroke (e.g. arteritis, dissection, migraine/vasospasm, drug misuse). Major risk sources of cardioembolism include permanent or paroxysmal atrial fibrillation, sustained atrial flutter, intracardiac thrombus, prosthetic cardiac valve, atrial myxoma or other cardiac tumours, mitral stenosis, recent (<4 weeks) myocardial infarction, left ventricular ejection fraction less than 30%, valvular vegetations, or infective endocarditis.

Recently, our group presented a descriptive analysis of an ESUS population derived from the Athens Stroke Registry. Among the overall ischemic stroke population, 10% of patients were classified as ESUS. These strokes were of mild-moderate severity and covert AF was identified as the underlying etiopathogenetic mechanism in approximately 40% of ESUS patients. The mortality risk in ESUS patients is lower compared to patients with cardioembolic stroke despite similar rates of stroke recurrence.

Also, the risk of stroke recurrence is higher in ESUS patients than in patients with non-cardioembolic strokes which could be a sign that the current antithrombotic strategy of treating ESUS patients with antiplatelets is suboptimal. Indeed, currently, it is not clear whether antiplatelets or anticoagulants are the ideal antithrombotic strategy in ESUS. Recently, two international, phase III, double-blind, randomized, controlled clinical trial were launched aiming to investigate whether anticoagulant treatment is superior to antiplatelet treatment for the secondary prevention in ESUS patient : the Randomized Evaluation in Secondary stroke Prevention Comparing the Thrombin inhibitor dabigatran etexilate versus aspirin in Embolic Stroke of Undetermined Source (RE-SPECT ESUS) trial and the NAVIGATE trial will compare dabigatran etexilate and rivaroxaban respectively to aspirin in ESUS patients.

It would be clinically useful to identify the predictors of covert AF in the ESUS population as this could possibly influence the choice of antithrombotic treatment, e.g. anticoagulants in ESUS patients at high risk of covert AF, and antiplatelets for ESUS patients with low risk of covert AF.

ELIGIBILITY:
Inclusion Criteria:

* 1. Embolic stroke of undetermined source (ESUS) defined as:

  * Ischemic stroke (including transient ischemic attack with positive neuroimaging) visualized by brain CT or MRI that is not lacunar (i.e., subcortical infarct ≤1.5 cm), and
  * Absence of cervical carotid atherosclerotic stenosis (or vertebral and basilar artery stenosis in case of posterior circulation stroke), that is ≥ 50%, or occlusion in arteries supplying the area of ischemia in CT or magnetic resonance (MR) angiography or ultrasound, and
  * No history of AF, no documented AF on 12-lead electrocardiogram (ECG) or episode of AF lasting 6 minutes or longer detected after ≥ 24-hour cardiac rhythm monitoring (Holter or telemetry), and
  * No intra-cardiac thrombus on transthoracic echocardiography, and
  * No other specific cause of stroke identified by routine clinical care (e.g., arteritis, dissection, migraine/vasospasm, drug abuse)
* 2. Age ≥18 years
* 3. Written informed consent

Exclusion Criteria:

* 1. ≥ 50% luminal stenosis or occlusion in arteries supplying the area of ischemia
* 2. History of AF
* 3. Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The dataset will be derived mainly from three high quality, prospective stroke registries: the Acute STroke Registry and Analysis of Lausanne (ASTRAL), the Athens Stroke Registry and the Larissa Stroke Outcome Registry (LASTRO)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | Twelve months
  Occurrence of atrial fibrillation during follow-up assessed either by 12-lead electrocardiogram (ECG) or telemetry or 24-hours Holter ECG, or longer-term ECG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: George Ntaios, MD, PhD, Principal Investigator — Medical School, University of Thessaly, Larissa University Hospital
Locations (3):
- Greece (2):
  - Department of Clinical Therapeutics, University of Athens, Alexandra Hospital, Athens
  - Medical School, University of Thessaly, Larissa University Hospital, Larissa
- Centre Cérébrovasculaire, Service de Neurologie, Département des Neurosciences Cliniques, Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hart RG, Diener HC, Coutts SB, Easton JD, Granger CB, O'Donnell MJ, Sacco RL, Connolly SJ; Cryptogenic Stroke/ESUS International Working Group. Embolic strokes of undetermined source: the case for a new clinical construct. Lancet Neurol. 2014 Apr;13(4):429-38. doi: 10.1016/S1474-4422(13)70310-7. PMID 24646875
- [Background] Ntaios G, Papavasileiou V, Milionis H, Makaritsis K, Vemmou A, Koroboki E, Manios E, Spengos K, Michel P, Vemmos K. Embolic Strokes of Undetermined Source in the Athens Stroke Registry: An Outcome Analysis. Stroke. 2015 Aug;46(8):2087-93. doi: 10.1161/STROKEAHA.115.009334. Epub 2015 Jul 9. PMID 26159795
- [Background] Ntaios G, Papavasileiou V, Milionis H, Makaritsis K, Manios E, Spengos K, Michel P, Vemmos K. Embolic strokes of undetermined source in the Athens stroke registry: a descriptive analysis. Stroke. 2015 Jan;46(1):176-81. doi: 10.1161/STROKEAHA.114.007240. Epub 2014 Nov 6. PMID 25378429
- [Background] Diener HC, Easton JD, Granger CB, Cronin L, Duffy C, Cotton D, Brueckmann M, Sacco RL; RE-SPECT ESUS Investigators. Design of Randomized, double-blind, Evaluation in secondary Stroke Prevention comparing the EfficaCy and safety of the oral Thrombin inhibitor dabigatran etexilate vs. acetylsalicylic acid in patients with Embolic Stroke of Undetermined Source (RE-SPECT ESUS). Int J Stroke. 2015 Dec;10(8):1309-12. doi: 10.1111/ijs.12630. Epub 2015 Sep 30. PMID 26420134
- [Derived] Kitsiou A, Sagris D, Schabitz WR, Ntaios G. Validation of the AF-ESUS score to identify patients with embolic stroke of undetermined source and low risk of device-detected atrial fibrillation. Eur J Intern Med. 2021 Jul;89:135-136. doi: 10.1016/j.ejim.2021.04.003. Epub 2021 May 2. No abstract available. PMID 33952425
- [Derived] Ntaios G, Weng SF, Perlepe K, Akyea R, Condon L, Lambrou D, Sirimarco G, Strambo D, Eskandari A, Karagkiozi E, Vemmou A, Korompoki E, Manios E, Makaritsis K, Vemmos K, Michel P. Data-driven machine-learning analysis of potential embolic sources in embolic stroke of undetermined source. Eur J Neurol. 2021 Jan;28(1):192-201. doi: 10.1111/ene.14524. Epub 2020 Oct 7. PMID 32918305
- [Derived] Ntaios G, Perlepe K, Lambrou D, Sirimarco G, Strambo D, Eskandari A, Karagkiozi E, Vemmou A, Korompoki E, Manios E, Makaritsis K, Vemmos K, Michel P. Identification of patients with embolic stroke of undetermined source and low risk of new incident atrial fibrillation: The AF-ESUS score. Int J Stroke. 2021 Jan;16(1):29-38. doi: 10.1177/1747493020925281. Epub 2020 May 19. PMID 32423317
- [Derived] Leventis I, Perlepe K, Sagris D, Sirimarco G, Strambo D, Georgiopoulos G, Eskandari A, Karagkiozi E, Vemmou A, Koroboki E, Manios E, Makaritsis K, Vemmos K, Michel P, Ntaios G. Characteristics and outcomes of Embolic Stroke of Undetermined Source according to stroke severity. Int J Stroke. 2020 Oct;15(8):866-871. doi: 10.1177/1747493020909546. Epub 2020 Mar 2. PMID 32122289
- [Derived] Perlepe K, Sirimarco G, Strambo D, Eskandari A, Karagkiozi E, Vemmou A, Koroboki E, Manios E, Makaritsis K, Vemmos K, Michel P, Ntaios G. Left atrial diameter thresholds and new incident atrial fibrillation in embolic stroke of undetermined source. Eur J Intern Med. 2020 May;75:30-34. doi: 10.1016/j.ejim.2020.01.002. Epub 2020 Jan 15. PMID 31952983
- [Derived] Ntaios G, Perlepe K, Lambrou D, Sirimarco G, Strambo D, Eskandari A, Karagkiozi E, Vemmou A, Koroboki E, Manios E, Makaritsis K, Vemmos K, Michel P. Prevalence and Overlap of Potential Embolic Sources in Patients With Embolic Stroke of Undetermined Source. J Am Heart Assoc. 2019 Aug 6;8(15):e012858. doi: 10.1161/JAHA.119.012858. Epub 2019 Jul 31. PMID 31364451
- [Derived] Ntaios G, Perlepe K, Sirimarco G, Strambo D, Eskandari A, Karagkiozi E, Vemmou A, Koroboki E, Manios E, Makaritsis K, Michel P, Vemmos K. Carotid plaques and detection of atrial fibrillation in embolic stroke of undetermined source. Neurology. 2019 Jun 4;92(23):e2644-e2652. doi: 10.1212/WNL.0000000000007611. Epub 2019 May 8. PMID 31068479